CLINICAL TRIAL: NCT02371044
Title: Point-of-Care Testing of Coagulation in Patients Treated With Direct Oral Anticoagulants 1
Acronym: POCT-DOAC 1
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Heart and Diabetes Center North Rhine-Westphalia (Other)
Responsible Party: Sponsor
Other Study IDs: .0 259/2013BO1
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Anticoagulation With Direct Oral Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples and citrated plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Rivaroxaban: N=20
- Apixaban: N=20
- Dabigatran: N=20

SUMMARY:
The investigators study aims to test the correlation between the CoaguChek point-of-care testing (POCT) device (Roche, Switzerland) and low plasma levels of all three currently approved direct oral anticoagulants (DOAC; rivaroxaban, apixaban and dabigatran) and to determine the diagnostic accuracy of POCT to rule out or detect relevant levels of DOAC in real-life stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients, who were newly started on oral anticoagulation with rivaroxaban, apixaban or dabigatran for secondary prevention of thromboembolic events
* Age ≥ 18 years

Exclusion Criteria:

* Vitamin K antagonists or direct oral anticoagulants ≤ 14 days prior to study participation
* Low-molecular weight heparin ≤ 24 hours
* Unfractionated heparin ≤ 12 hours
* Abnormal coagulation values at baseline (Quick < 70% or activated thromboplastin time (aPTT) > 40sec.)
* History of coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive stroke patients, who were newly started on oral anticoagulation with rivaroxaban, apixaban or dabigatran for secondary prevention of thromboembolic events.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Effect/Correlation of direct oral anticoagulants (DOAC) on CoaguChek point-of-care testing (POCT) result | 24 hours
  DOAC concentrations determined by ultra-performance liquid chromatography-tandem mass spectrometry

SECONDARY OUTCOMES:
Diagnostic accuracy of the CoaguChek POCT to rule out or detect relevant DOAC levels | 24h
Effect/Correlation of DOAC on prothrombin time (PT), activated thromboplastin time (aPTT), anti-Xa activity and Hemoclot assay | 24h

CONTACTS AND LOCATIONS:
Overall Officials: Sven Poli, Dr., Principal Investigator — University Hospital Tuebingen

REFERENCES:
- [Derived] Ebner M, Birschmann I, Peter A, Hartig F, Spencer C, Kuhn J, Blumenstock G, Zuern CS, Ziemann U, Poli S. Emergency Coagulation Assessment During Treatment With Direct Oral Anticoagulants: Limitations and Solutions. Stroke. 2017 Sep;48(9):2457-2463. doi: 10.1161/STROKEAHA.117.017981. Epub 2017 Aug 3. PMID 28775134
- [Derived] Ebner M, Peter A, Spencer C, Hartig F, Birschmann I, Kuhn J, Wolf M, Winter N, Russo F, Zuern CS, Blumenstock G, Ziemann U, Poli S. Point-of-Care Testing of Coagulation in Patients Treated With Non-Vitamin K Antagonist Oral Anticoagulants. Stroke. 2015 Oct;46(10):2741-7. doi: 10.1161/STROKEAHA.115.010148. Epub 2015 Aug 13. PMID 26272385